CLINICAL TRIAL: NCT01711528
Title: Phase 1 Clinical Trial of a Novel CDK Inhibitor Dinaciclib (SCH 727965) in Combination With Bortezomib and Dexamethasone in Relapsed Multiple Myeloma
Brief Title: Dinaciclib, Bortezomib, and Dexamethasone in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01737; NCI-2012-01737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1113; NCI 9157; CDR0000741989; MC1113 (Other: Mayo Clinic); 9157 (Other: CTEP); P30CA015083 (NIH); R01CA167511 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH); UM1CA186716 (NIH); NCT02668731 (obsolete NCT alias)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; dinaciclib

ARMS (2):
- Schedule I (dinaciclib, bortezomib, dexamethasone) (Experimental): Patients receive dinaciclib IV over 2 hours and bortezomib SC or IV (if patients do not tolerate SC injection) on days 1, 8, and 15 and dexamethasone PO QD on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Dinaciclib; Other: Laboratory Biomarker Analysis
- Schedule II (dinaciclib, bortezomib, dexamethasone) (Experimental): Patients receive dinaciclib IV over 2 hours on day 1; bortezomib SC on days 1 and 8; and dexamethasone PO QD on days 1, 2, 8, and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Dinaciclib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Dinaciclib — Given IV
  Other Names: CDK Inhibitor SCH 727965; MK-7965; SCH 727965
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of dinaciclib and bortezomib when given together with dexamethasone in treating patients with multiple myeloma that has returned after a period of improvement. Dinaciclib and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving dinaciclib and bortezomib together with dexamethasone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated doses of dinaciclib and bortezomib, when used in combination, in two different schedules, for treatment of relapsed multiple myeloma.

SECONDARY OBJECTIVES:

I. To determine the toxicities associated with dinaciclib and bortezomib, when used in combination, for treatment of relapsed multiple myeloma.

II. To determine the overall response rate associated with dinaciclib and bortezomib, when used in combination, for treatment of relapsed multiple myeloma.

III. To explore the differences in toxicity associated with two different schedules of dinaciclib and bortezomib used in combination.

TERTIARY OBJECTIVES:

I. To examine if expression levels of target cyclin dependent kinase (CDK): CDK 2,5,7 and 9 levels in cluster of differentiation (CD)138-purified tumor cells, will be correlated with response (clinical and molecular) to determine if high or low level target CDK expression, if present, influences dinaciclib efficacy.

II. To examine if immunoglobulin (Ig)H translocation status, P53 status and presence of v-myc myelocytomatosis viral oncogene homolog (avian) (Myc) amplification or rearrangement, determined on patient bone marrow before treatment, using a pre validated fluorescence in situ hybridization (FISH) panel to identify common myeloma translocations, will be correlated with molecular and/or clinical markers of drug activity, and to assess if specific genetic subgroups of myeloma tumors are responsive or resistant.

III. To determine the gene expression profiles of myeloma cells before and after treatment to understand the role of tumor gene dysregulation and/or dinaciclib induced effects on transcription.

OUTLINE: This is a dose-escalation study of dinaciclib and bortezomib. Patients are assigned to 1 of 2 treatment schedules.

SCHEDULE I: Patients receive dinaciclib intravenously (IV) over 2 hours and bortezomib subcutaneously (SC) or IV (if patients do not tolerate SC injection) on days 1, 8, and 15 and dexamethasone orally (PO) once daily (QD) on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

SCHEDULE II: Patients receive dinaciclib IV over 2 hours on day 1; bortezomib SC on days 1 and 8; and dexamethasone PO QD on days 1, 2, 8, and 9. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine =< 2.5 mg/dL
* Absolute neutrophil count >= 1000/uL
* Untransfused platelet count >= 75000/uL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
* Patients with relapsed multiple myeloma who have already received one or more standard treatment regimens
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Adequate residual organ function per treating physician discretion; Note: there is no limit with regard to the number of prior therapies
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to provide samples for correlative research purposes
* Willing to return to consenting institution for follow-up during the study
* Recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior antineoplastic therapy

Exclusion Criteria:

* Any of the following recent therapies:

  * Alkylators (e.g. melphalan, cyclophosphamide) =< 14 days prior to registration
  * Anthracyclines =< 14 days prior to registration
  * High dose corticosteroids, immune modulatory drugs (thalidomide or lenalidomide), or proteosome inhibitors (bortezomib) =< 7 days prior to registration
* Concomitant high dose corticosteroids (concurrent use of corticosteroids); EXCEPTION: patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than amyloid, i.e., adrenal insufficiency, rheumatoid arthritis, etc.
* Other active malignancy =< 2 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of study drug
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 30 days after stopping treatment
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 2 on clinical examination during the screening period
* Major surgery =< 14 days prior to registration
* Currently taking strong or moderate inhibitors/inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); Note: dinaciclib is a CYP3A4 substrate; patients should not take grapefruit/grapefruit juice or St. John's wort; use of strong or moderate CYP3A4 inhibitors is prohibited from < 7 days prior to registration; use of CYP3A4 inducers is prohibited from =< 7 days prior to registration
* Any of the following conditions:

  * Myocardial infarction =< 6 months prior to registration or has New York Heart Association (NYHA) class III or IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Electrocardiographic evidence of acute ischemia
  * Active conduction system abnormalities; NOTE: prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Known hypersensitivity to bortezomib, boron, or mannitol
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study per the judgment of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
MTD of dinaciclib and bortezomib when given together with dexamethasone, based on the incidence of dose-limiting toxicity (DLT), graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 28 days
  MTD is defined as the dose level below the lowest dose that induces DLT in at least one-third of patients.

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to NCT CTCAE version 4.0 | Up to 3 months
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. Toxicity is defined as adverse events that are classified as possibly, probably, or definitely related to study treatment. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Overall response rate | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time to progression | Up to 3 months
  Summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patients, assessed up to 3 months
  Summarized descriptively.
Time until hematologic nadirs (absolute neutrophil count, platelets, hemoglobin) | Up to 3 months
  Summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin